CLINICAL TRIAL: NCT00157079
Title: A Clinical Investigation to Assess the Safety and Efficacy of Immune Globulin Intravenous (Human), 10% in Subjects With Primary Immunodeficiency Disorders
Brief Title: Safety and Efficacy Study of a 10% Intravenous Immune Globulin Solution in Subjects With Primary Immunodeficiency Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: 160101
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Primary Immunodeficiency Diseases (PID); Immune Thrombocytopenic Purpura (ITP); Kawasaki Syndrome
Keywords: PID; Immunodeficiency; Immune Thrombocytopenic Purpura (ITP); Kawasaki syndrome
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Purpura, Thrombocytopenic, Idiopathic; Mucocutaneous Lymph Node Syndrome; Immunologic Deficiency Syndromes | interventions — gamma-Globulins

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

INTERVENTIONS:
Biological: Immune Globulin Intravenous (Human), 10%

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Immune Globulin Intravenous (Human), 10% (IGIV 10%) in subjects with primary immunodeficiency disorders.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from either the subject or the subject's legally acceptable representative prior to any study-related procedures and study product administration
* Diagnosis of a PID disorder as defined by World Health Organization criteria for which the subject has been receiving a regimen of IGIV infusions every 21 to 28 days over a period of at least 4 months pre-study at a dose of 300-600 mg/kg body weight
* Subjects > 24 months of age
* A negative serum pregnancy test for any female subject who is of childbearing potential.

Exclusion Criteria:

* Subjects sero-positive at enrollment for one or more of the following: hepatitis B surface antigen (HBsAg), antibodies to hepatitis C virus (HCV), antibodies to human immunodeficiency virus (HIV) Types 1 or 2
* Subjects with levels of alanine amino transferase (ALT) and aspartate amino transferase (AST) > 2.5 times the upper limit of normal for the testing laboratory. An AST > 2.5 times the upper limit of normal is allowable, if the ALT does not exceed the upper limit of the reference range for the testing laboratory
* Subjects with neutropenia (defined as an ANC >= 1,000/mm3)
* Subjects with serum creatinine levels greater than two times the upper limit of normal for age and gender
* Subjects with malignancy or a history of malignancy
* Subjects who received any blood or blood product exposure other than an IGIV and/or immune serum globulin (ISG) preparation within the 6 months prior to study entry
* Subjects with an ongoing history of hypersensitivity or persistent reactions (urticaria, breathing difficulty, severe hypotension, or anaphylaxis) following IGIV and/or ISG infusions
* Subjects with selective complete IgA deficiency
* Subjects with moderate levels of anti-IgA antibodies (>150), or subjects with lower anti-IgA antibodies who are naive to IGIV treatment. (Subjects with lower levels of IgA antibodies, whom the investigators know to have tolerated IgA containing IGIV preparations in the past, may be included if the investigator is comfortable with this)
* Subjects receiving antibiotic therapy for the treatment of infection within 30 days prior to enrollment
* Subjects who receive prophylactic antibiotics as part of their care regimen
* Subjects participating in another clinical study involving an investigational product or device within 30 days prior to study entry

Min Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2002-06-25 (Actual); Primary Completion 2003-12-16 (Actual); Study Completion 2003-12-16 (Actual)

PRIMARY OUTCOMES:
Mean number of acute serious bacterial infections per participant per year | Throughout the study period of 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (11):
- United States (11):
  - Children´s Hospital Los Angeles, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - 1st Allergy and Clinical Research Center, Englewood, Colorado
  - Allergy Associates of the Palm Beaches, North Palm Beach, Florida
  - University of South Florida; Asthma, Allergy & Immunology CRU, Tampa, Florida
  - Rush Presbyterian - St. Lukes Medical Center, Chicago, Illinois
  - Children´s Hospital Boston, Boston, Massachusetts
  - Allergy, Asthma & Immunology Assoc., Omaha, Nebraska
  - Asthma and Allergy Center, Papillion, Nebraska
  - Montefiore Medical Center, Albert Einstein College of Medicine, The Bronx, New York
  - Pediatric Allergy/Immunology Associates, Dallas, Texas